CLINICAL TRIAL: NCT04899960
Title: Drug-Related Problems in Neonatal Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nadir Yalçın, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA-20004
Record Dates: First submitted 2021-05-11; First posted 2021-05-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-05

CONDITIONS: Neonatal Intensive Care Unit; Medication Errors; Drug-Related Problems; Adverse Drug Event; Drug-Drug Interaction; Clinical Pharmacy; Machine Learning
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Observational Group (No Intervention)
- Control (Validation) Group (No Intervention)
- İnterventional Group (Experimental)
  Interventions: Drug: Clinical Pharmacist Intervention

INTERVENTIONS:
Drug: Clinical Pharmacist Intervention — Prevention of drug-related problems by clinical pharmacist in neonatal intensive care unit.
  Arms: İnterventional Group

SUMMARY:
Drug-related problems in newborn babies have been reported with a rate of 4-30%. It is estimated that the higher rates of these problems in hospitalized children under the age of two are related to the variety of drugs used and the differences in the age, weight and diagnosis of the patients. In this context, with the clinical parameters and demographic data obtained in the first 24 hours of the patients hospitalized in the neonatal intensive care unit, machine learning algorithms are used to predict the risks that may arise from possible drug-related problems (prescribing and administration errors, side effects and drug-drug interactions) that may occur during hospitalization. The algorithm, which will be created by modeling with a high number of big data pool, is planned to be transformed into a clinical decision support system software that can be used easily in clinical practice with online and mobile applications. By processing the data of the patients to be included in the model, it is aimed to prevent and manage drug-related problems before they occur, as well as to provide cost-effective medşcation treatment to patients hospitalized in the neonatal intensive care unit, together with a reduction in the risk of drug-related mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Newborns aged 0-28 days,
* Consent form taken by the parents to participate in the study,
* Patients admitted to neonatal intensive care unit or surgical wards

Exclusion Criteria:

* Have a postnatal age greater than 28 days,
* Patients who will not be given any medication,
* Patients who took part in any drug research within the last 28 days

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 512 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Score for Neonatal Acute Physiology and Perinatal Extension Score | Through study completion, an average of 1 year.
  Score for Neonatal Acute Physiology and Perinatal Extension Score is predictor of mortality in neonates.
Neonatal Therapeutic Intervention Scoring System | Through study completion, an average of 1 year.
  It is a therapy-based severity of illness (morbidity) assessment index.
Neonatal Early-Onset Sepsis Risk Score | Through study completion, an average of 1 year.
  It is use first week of life for determined sepsis risk with gestational age, highest maternal antepartum temperature, duration of rupture of membranes, etc.
Neonatal Nutrition Screening Tool | Through study completion, an average of 1 year.
  It could be used on all infants in the neonatal intensive care on a weekly basis by nursing staff to identify those at high risk of poor growth and in need of additional nutrition support during their stay.

SECONDARY OUTCOMES:
Neonatal Adverse Event Severity Scale | Through study completion, an average of 1 year.
  It describes a consensus process that led to the development of standard severity criteria for neonatal adverse events. The use of this tool could improve the quality of drug and device safety evaluations and facilitate the conduct of neonatal clinical trials.
The Drug Interaction Probability Scale | Through study completion, an average of 1 year.
  This scale uses a series of questions relating to the potential drug interaction to estimate a probability score.
Adverse Drug Reactions Algorithm for Infants | Through study completion, an average of 1 year.
  The new algorithm developed using actual patient data is more valid and reliable than the Naranjo algorithm for identifying adverse drug reactions in the neonatal intensive care unit population.
National Aeronautics and Space Administration Task Load Index | Through study completion, an average of 1 year.
  NASA Task Load Index (NASA-TLX) is a widely used, subjective, multidimensional assessment tool that rates perceived workload in order to assess a task, system, or team's effectiveness or other aspects of performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Yalçın, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Nadir Yalçın, Ankara, TR, Turkey (Türkiye)

REFERENCES:
- [Derived] Yalcin N, Kasikci M, Celik HT, Allegaert K, Demirkan K, Yigit S. Impact of clinical pharmacist-led intervention for drug-related problems in neonatal intensive care unit a randomized controlled trial. Front Pharmacol. 2023 Aug 14;14:1242779. doi: 10.3389/fphar.2023.1242779. eCollection 2023. PMID 37645440
- [Derived] Yalcin N, Kasikci M, Celik HT, Allegaert K, Demirkan K, Yigit S, Yurdakok M. Development and validation of a machine learning-based detection system to improve precision screening for medication errors in the neonatal intensive care unit. Front Pharmacol. 2023 Apr 14;14:1151560. doi: 10.3389/fphar.2023.1151560. eCollection 2023. PMID 37124199